CLINICAL TRIAL: NCT01031771
Title: Clinical and Instrumental Evaluation of Swallowing in Children With Cerebral Palsy
Acronym: CP
Status: Completed | Type: Observational
Sponsor: Fortaleza University (Other)
Responsible Party: Moisés Andrade dos Santos de Queiroz, Fortaleza University
Other Study IDs: 105/09
Record Dates: First submitted 2009-12-12; First posted 2009-12-15 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2009-12

CONDITIONS: Cerebral Palsy; Deglutition Disorders
Keywords: Cerebral Palsy; Deglutition; Deglutition disorders; Endoscopy
MeSH Terms: conditions — Cerebral Palsy; Deglutition Disorders

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to correlate the alimentary consistencies and deglutition disorders in children with cerebral palsy.

DETAILED DESCRIPTION:
Cross-sectional and quantitative study with sample consisted of 50 children with cerebral palsy. The data collection consisted in detection of the main dysphagic manifestations in different consistency of food and types of cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Children with Cerebral Palsy diagnoses were involved, independent from the pre, peri and postnatal factors and from the type of Cerebral Palsy

Exclusion Criteria:

* Children who presented oropharyngelarynx structural abnormality and/or impossibility to feed by oral way

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with Cerebral Palsy diagnoses
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-02; Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Moisés A Queiroz, Graduate, Principal Investigator — Fortaleza University